CLINICAL TRIAL: NCT00817778
Title: A Randomised, Single-Blind, Placebo-Controlled, Phase IIA Study to Assess the Safety and Tolerability After Multiple Oral Doses of AZD1656 in Patients With Type 2 Diabetes Mellitus Treated With Metformin
Brief Title: Study to Assess the Safety and Tolerability After Multiple Oral Doses of AZD1656 in Patients With Type 2 Diabetes Mellitus Treated With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00019
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes
Keywords: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1656 (Experimental): Dose titration of oral suspension during 4 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 24 days
  Interventions: Drug: AZD1656
- Placebo (Placebo Comparator): Dose titration of oral suspension during 4 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 24 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Subjects will be treated with tolerable dose twice daily for another 24 days.
  Arms: AZD1656
Drug: Placebo — Subjects will be treated with tolerable dose twice daily for another 24 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the 1 month safety and tolerability after multiple oral doses of AZD1656 in patients with Type 2 Diabetes Mellitus Treated with Metformin

ELIGIBILITY:
Inclusion Criteria:

* Male or women of non-childbearing potential (postmenopausal, and/or have undergone hysterectomy and/or bilateral oophorectomy or salpingectomy/ tubal ligation)
* Ongoing treatment with metformin on a stable dose of ≥ 1500 mg/day for at least 8 weeks prior to randomisation
* HbA1c ≤ 10% at enrolment (HbA1c value according to international Diabetes Control and Complications Trial [DCCT] standard)

Exclusion Criteria:

* History of ischemic heart disease, symptomatic heart failure, stroke, transitory ischemic attack or symptomatic peripheral vascular disease
* Clinically significant abnormalities in ECG, clinical chemistry, haematology, or urine analysis results. Positive test for Hepatitis B surface antigen or antibodies to human immunodeficiency virus (HIV) or antibodies to Hepatitis C virus

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof, Study Director — AstraZeneca R&D Mölndal; Emanuel P DeNoia, M.D, Principal Investigator — Healthcare Discoveries LLC Icon Development Solutions
Locations (1):
- Research Site, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: AZD1656
- Placebo Comparator: Placebo
Period: Overall Study
Arm/Group | Experimental | Placebo Comparator
Started | 19 | 8
Completed | 16 | 5
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Study-specific discontinuation criteria | 0 | 1
Not completed — Poor venous access | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo Comparator | Total
Number analyzed (Participants) | 19 | 8 | 27
Age Continuous [Mean (Full Range); unit: years] | 60.2 [39 to 72] | 60.3 [34 to 74] | 60.2 [34 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure, Change From Baseline to End of Treatment
Time Frame: Baseline is pre-dose first day of dosing, end of treatment is the morning following the treatment period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
mmHg | -0.5 (11.48) | 9.2 (10.43)

2. Primary Outcome: Diastolic Blood Pressure, Change From Baseline to End of Treatment
Time Frame: Baseline is pre-dose first day of dosing, end of treatment is the morning following the treatment period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
mmHg | -0.2 (6.20) | 2.0 (10.32)

3. Primary Outcome: Pulse, Change From Baseline to End of Treatment
Time Frame: Baseline is pre-dose first day of dosing, end of treatment is the morning following the treatment period
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
beats/min | 2.7 (5.69) | -1.6 (6.23)

4. Primary Outcome: Weight, Change From Baseline to End of Treatment
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
kg | 0.2 (1.00) | 0.0 (3.81)

5. Primary Outcome: Clinically Relevant Change of Laboratory Variables
Description: Number of participants with clinically relevant change of laboratory variables (clinical chemistry, haematology and urinalysis parameters
Time Frame: Measured regularly from day before first dose to day after last dose
Measure: Number; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 19 | 8
Participants | 0 | 0

6. Secondary Outcome: Area Under the Plasma Concentration vs Time Curve (AUC0-24) of AZD1656
Description: Dose-adjusted to a total daily dose of 100 mg due to titrated doses
Time Frame: Measured last day of treatment
Measure: Geometric Mean (Standard Deviation); unit: umol*h/L
Arm/Group | Experimental
Number analyzed (Participants) | 16
umol*h/L | 23.17 (7.46)

7. Secondary Outcome: Maximum Plasma Concentration of AZD1656
Description: Dose-adjusted to a morning dose of 50 mg due to titrated doses
Time Frame: Measured last day of treatment
Measure: Geometric Mean (Standard Deviation); unit: umol/L
Arm/Group | Experimental
Number analyzed (Participants) | 16
umol/L | 1.90 (0.99)

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration of AZD1656
Time Frame: Measured last day of treatment
Measure: Median (Full Range); unit: h
Arm/Group | Experimental
Number analyzed (Participants) | 16
h | 0.625 [0.25 to 6.00]

9. Secondary Outcome: Terminal Elimination Half-life of AZD1656
Time Frame: Measured following the afternoon dose last day of treatment
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | Experimental
Number analyzed (Participants) | 10
h | 7.07 [2.48 to 12.93]

10. Secondary Outcome: Apparent Oral Clearance of AZD1656
Time Frame: Measured last day of treatment
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | Experimental
Number analyzed (Participants) | 16
L/h | 9.02 [5.39 to 13.94]

11. Secondary Outcome: P-Glucose (AUC0-24)/24, Change From Baseline to End of Treatment
Description: Log ratio (End of treatment/Baseline) has been analysed in a mixed-effect ANOVA model, using treatment as fixed effect and log(Baseline) as covariate. Resulting estimates have been back-transformed from the log-scale and then multiplied by 100 to obtain the relative ratio (end of treatment/placebo) in percent.
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Relative ratio in percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
Relative ratio in percent | 75.85 [69.82 to 82.39] | 99.42 [85.05 to 116.23]

12. Secondary Outcome: S-Insulin (AUC0-24)/24, Change From Baseline to End of Treatment
Description: as for outcome 11
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Relative ratio in percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
Relative ratio in percent | 103.81 [90.75 to 118.74] | 86.06 [67.24 to 110.14]

13. Secondary Outcome: S-C-Peptide (AUC0-24)/24, Change From Baseline to End of Treatment
Description: as for outcome 11
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Relative ratio in percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 16 | 5
Relative ratio in percent | 103.60 [97.10 to 110.54] | 98.01 [87.10 to 110.29]

ADVERSE EVENTS:
Arm/Group | Experimental | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/8
Other Adverse Events (participants affected / at risk) | 15/19 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=19) | Placebo Comparator (N=8)
Rapid Atrial Fibrillation (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=19) | Placebo Comparator (N=8)
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood Glucose Decreased (Injury, poisoning and procedural complications) | 9 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 2
Tremor (Nervous system disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The primary objective of the study was to assess safety and tolerability and hence the study was not sized based on statistical considerations. The most import outcome, "no safety or tolerability concerns were identified", is not a numerical variable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CONTRACT RESEARCH ORGANIZATION AGREEMENT by and between ASTRAZENECA AB and the CRO. CRO agrees that AstraZeneca shall have the exclusive right to publish the results of the Study, including all Work Product, and that such results may not be published or otherwise disseminated by CRO without the prior written approval of AstraZeneca.